CLINICAL TRIAL: NCT04566653
Title: Non-Interventional, Exploratory, Phase IV, Single-Blind, Cross-Sectional, Randomised, Cross-over Study Evaluating Patient Palatability and Preference of 3 Potassium Binders in Patients With Chronic Kidney Disease & Hyperkalaemia (APPETIZE).
Brief Title: Patient Palatability and Preference of 3 Potassium Binders in Patients With Chronic Kidney Disease and Hyperkalaemia
Acronym: APPETIZE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry); Calyx (Unknown); ERT: Clinical Trial Technology Solutions (Other); Medidata Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480C00016
Record Dates: First submitted 2020-07-31; First posted 2020-09-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Disease + Hyperkalaemia +/- Heart Failure
Keywords: palatability; Lokelma; hyperkalaemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia | interventions — polystyrene sulfonic acid; Water; sodium zirconium cyclosilicate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dialysis-dependent: chronic kidney disease patients with hyperkalaemia and dialysis-dependent
  Interventions: Drug: Calcium Polystyrene Sulphonate 15g/60 mL water; Drug: Lokelma® 5 g/45mL water; Drug: Veltassa® 8,4 g/80mL water; Drug: Sodium Polystyrene Sulphonate 15g/60 mL water
- non-dialysis-dependent: chronic kidney disease patients with hyperkalaemia and non-dialysis-dependent
  Interventions: Drug: Calcium Polystyrene Sulphonate 15g/60 mL water; Drug: Lokelma® 10 g/45 mL water; Drug: Veltassa® 8,4 g/80mL water; Drug: Sodium Polystyrene Sulphonate 15g/60 mL water

INTERVENTIONS:
Drug: Calcium Polystyrene Sulphonate 15g/60 mL water — K+ binder, not for treatment but for tasting (sip-and-spit taste test)
Drug: Lokelma® 5 g/45mL water — K+ binder, not for treatment but for tasting (sip-and-spit taste test)
  Groups: dialysis-dependent
Drug: Lokelma® 10 g/45 mL water — K+ binder, not for treatment but for tasting (sip-and-spit taste test)
  Groups: non-dialysis-dependent
Drug: Veltassa® 8,4 g/80mL water — K+ binder, not for treatment but for tasting (sip-and-spit taste test)
Drug: Sodium Polystyrene Sulphonate 15g/60 mL water — K+ binder, not for treatment but for tasting (sip-and-spit taste test)

SUMMARY:
This non-interventional, Phase IV, exploratory, cross-over, randomised, single-blind, active comparator-controlled study has been designed to measure the palatability and preference of Lokelma® versus Veltassa® versus S/CPS in patients with dialysis and non-dialysis chronic kidney disease (CKD) and hyperkalaemia (HK). The sponsor hypothesizes that palatability, in terms of taste, texture, smell, and mouthfeel, will score higher (better) for Lokelma when compared with Veltassa and S/CPS.

DETAILED DESCRIPTION:
This non-interventional, Phase IV, exploratory, cross-over, randomised, single-blind, active comparator-controlled study has been designed to measure the palatability and preference of sodium zirconium cyclosilicate (hereafter referred to as Lokelma®) versus calcium patiromer sorbitex (hereafter referred to as Veltassa®) versus sodium polystyrene sulphonate (SPS) or calcium polystyrene sulphonate (CPS) (hereafter referred to as S/CPS) in patients with dialysis and non-dialysis chronic kidney disease (CKD) and hyperkalaemia (HK). The sponsor hypothesizes that palatability, in terms of taste, texture, smell, and mouthfeel, will score higher (better) for Lokelma when compared with Veltassa and S/CPS. Each objective will be analysed per country. In addition, the difference in results per regions and overall may be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be adults aged ≥18 years, at the time of signing the informed consent.
2. Participants should have CKD defined by having an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (calculated using CKD-EPI equation) measured twice at least 90 days apart. (The eGFR should be measured when the participant is considered to be in a steady state without recent changes in volume status, medications that could impact the result (eg, nonsteroidal anti-inflammatory drugs, aminoglycosides, co-trimoxazole), or changes in dietary protein intake.)
3. Prevalent HK with serum K+ >5 mmol/L.
4. Male and/or female
5. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Informed consent must be obtained prior to any study-specific procedures performed.

Exclusion Criteria:

1. Screening serum K+ value which, in the opinion of the investigator, requires immediate medical intervention (ie, cannot wait until after tasting procedures).
2. As judged by the investigator, any evidence of any condition which in the investigator's opinion makes it undesirable for the participant to participate in the study.
3. Known history of drug or alcohol abuse within 6 months of screening.
4. History of QT prolongation associated with other medications that required discontinuation of that medication, including congenital long QT syndrome.
5. Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication are permitted.
6. Have a life expectancy of <6 months.
7. 12-lead ECG with reported QTcF >550 msec at screening.
8. Are current smoker.
9. Have mouth ulcers/mouth infection, respiratory infection, nasal congestion, or other condition, medication, or procedure which may interfere with sense of smell or taste, in opinion of the investigator.
10. Participants currently prescribed a K+ binder at time of screening/enrolment.
11. Participants unable to hold other oral medications from 3 hours prior to the start of tasting through 3 hours after the end of tasting.
12. Current participation or participation within the previous 28 days in another clinical study with an investigational product administered.
13. Participants with a known hypersensitivity to Lokelma, Veltassa, or S/CPS or any of the excipients of the NIMPs.
14. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
15. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
16. Previous enrolment or randomisation in the present study.
17. For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
18. Participants unable to read the local language and therefore unable to complete the questionnaires.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dialysis and non-dialysis CKD and HK
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Difference in scores (0-40) for overall palatability of NIMPs | Tasting visit (day 1)
  To compare patient-reported overall palatability (composite of taste, texture, smell, and mouthfeel) between Lokelma and Veltassa, and between Lokelma and S/CPS in the United States (US)

SECONDARY OUTCOMES:
Difference in scores (0-40) for overall palatability of NIMPs | Tasting visit (day 1)
  To compare patient-reported overall palatability (composite of taste, texture, smell, and mouthfeel) between Lokelma and Veltassa, and between Lokelma and S/CPS in Canada
Difference in scores (0-40) for overall palatability of NIMPs | Tasting visit (day 1)
  To compare patient-reported overall palatability (composite of taste, texture, smell, and mouthfeel) between Lokelma and Veltassa, and between Lokelma and S/CPS in the European Union (EU)
Difference in scores for feelings of Appeal (4-36), Engagement (4-36), and Empowerment (4-36) regarding taste overall palatability of NIMPs using the AdSAM emotional response tool | Tasting visit (day 1)
  To compare patient-reported emotional response to overall palatability (composite of taste, texture, smell, and mouthfeel) taste between Lokelma and Veltassa, and between Lokelma and S/CPS in the US
Difference in scores for feelings of appeal (4-36), engagement (4-36), and empowerment (4-36) regarding overall palatability of NIMPs using the AdSAM emotional response tool | Tasting visit (day 1)
  To compare patient-reported emotional response to overall palatability (composite of taste, texture, smell, and mouthfeel) between Lokelma and Veltassa, and between Lokelma and S/CPS in Canada
Difference in scores for feelings of appeal (4-36), engagement (4-36), and empowerment (4-36) regarding overall palatability of NIMPs using the AdSAM emotional response tool | Tasting visit (day 1)
  To compare patient-reported emotional response to overall palatability (composite of taste, texture, smell, and mouthfeel) between Lokelma and Veltassa, and ,between Lokelma and S/CPS in the EU
Scoring of palatability (0-40), Appeal of palatability (4-36), Engagement of palatability (4-36), Empowerment of palatability (4-36), Overall composite emotional strength indicator scores (0-1200), Feelings towards palatability | Tasting Visit (day 1)
  To describe patient-reported preference for overall palatability (composite of taste, texture, smell, and mouthfeel) (scoring and non-verbal emotional response for how each NIMP made patients feel ofto each NIMP) of 3 currently marketed K+ binders ((of Lokelma, Veltassa, and S/CPS) in the US, Canada, and EU, respectively)
Scoring (0-10), Appeal (9-1), Engagement (9-1), Empowerment (1-9), Overall emotional strength indicator score (0-300), and Feelings towards willingness to take a K+ binder | Tasting Visit (day 1)
  To describe and compare, based on the overall palatability experience, scoring and emotional response for how willing patients would be to take each K+ binder to help manage their serum potassium (likelihood of adherence) in the US, Canada, and EU
Overall preference ranking of NIMPs (1, 2, or 3) of Lokelma, Veltassa, and S/CPS • Use of Comparative AdSAM Emotional Strength Index and Emotional TempIndicator scores to derive overall preference | Tasting visit (day 1)
  To describe patient-reported preference by ranking the NIMPs, and derived preference based on the emotional strength indexindicator scores in the US, Canada, and EU

OTHER OUTCOMES:
See primary and secondary endpoints | Tasting visit (day 1)
  Overall palatability scores (0-40) between Lokelma and Veltassa, and between Lokelma and S/CPS will be described and compared for all primary and secondary endpoints for: North America, per individual EU countries (where data permit), and over all countries/regions
See primary and secondary endpoints | Tasting visit (day 1)
  Patient preference between Lokelma and Veltassa, and between Lokelma and S/CPS will be described and compared for all primary and secondary endpoints for: North America, per individual EU countries (where data permit), and over all countries/regions.
Categories or combinations based on Appeal of each attribute (taste, texture, smell, and mouthfeel) | Tasting visit (day 1)
  Appeal test score (1-9) for each attribute (taste, texture, smell, and mouthfeel) will be measured using AdSAM questionnaires using published research and analysed using AdSAM methodology and compare between Lokelma and Veltassa, and between Lokelma and S/CPS for the US, Canada, EU, North America, per individual EU countries (where data permit), and over all countries/regions.
Categories or combinations based on Engagement of each attribute (taste, texture, smell, and mouthfeel) | Tasting visit (day 1)
  Engagement test score (1-9) for each attribute (taste, texture, smell, and mouthfeel) will be measured using AdSAM questionnaires team using published research and analysed using AdSAM methodology and compare between Lokelma and Veltassa, and between Lokelma and S/CPS for the US, Canada, EU, North America, per individual EU countries (where data permit), and over all countries/regions
Categories or combinations based on Empowerment of each attribute (taste, texture, smell, and mouthfeel) | Tasting visit (day 1)
  Empowerment test score (1-9) for each attribute (taste, texture, smell, and mouthfeel) will be measured using AdSAM questionnaires team using published research and analysed using AdSAM methodology and compare between Lokelma and Veltassa, and between Lokelma and S/CPS for the US, Canada, EU, North America, per individual EU countries (where data permit), and over all countries/regions
Scoring (0-10) of taste, texture, smell, and mouthfeel | Tasting visit (day 1)
  Scores of individual palatability attributes (taste, texture, smell, and mouthfeel) will be described individually by countries/regions
Determining specific feelings regarding taste, texture, smell, and mouthfeel using the AdSAM emotional response model | Tasting visit (day 1)
  Emotional response of individual palatability attributes (taste, texture, smell, and mouthfeel) will be described individually by countries/regions

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wittbrodt, PharmD, MPH, Study Director — AstraZeneca, Biopharmaceuticals Medical
Locations (18):
- United States (2):
  - Research Site, Temple Terrace, Florida
  - Research Site, West Palm Beach, Florida
- Canada (4):
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (3):
  - Research Site, Amiens
  - Research Site, Boulogne-Billancourt
  - Research Site, Nice
- Italy (3):
  - Research Site, Genova
  - Research Site, Parma
  - Research Site, Pavia
- Spain (4):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
- Sweden (2):
  - Research Site, Eskilstuna
  - Research Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Thomsen RW, Nicolaisen SK, Hasvold P, Sanchez RG, Pedersen L, Adelborg K, Egstrup K, Egfjord M, Sorensen HT. Elevated potassium levels in patients with chronic kidney disease: occurrence, risk factors and clinical outcomes-a Danish population-based cohort study. Nephrol Dial Transplant. 2018 Sep 1;33(9):1610-1620. doi: 10.1093/ndt/gfx312. PMID 29177463
- [Background] Laureati P, Xu Y, Trevisan M, Schalin L, Mariani I, Bellocco R, Sood MM, Barany P, Sjolander A, Evans M, Carrero JJ. Initiation of sodium polystyrene sulphonate and the risk of gastrointestinal adverse events in advanced chronic kidney disease: a nationwide study. Nephrol Dial Transplant. 2020 Sep 1;35(9):1518-1526. doi: 10.1093/ndt/gfz150. PMID 31377791
- [Background] Noel JA, Bota SE, Petrcich W, Garg AX, Carrero JJ, Harel Z, Tangri N, Clark EG, Komenda P, Sood MM. Risk of Hospitalization for Serious Adverse Gastrointestinal Events Associated With Sodium Polystyrene Sulfonate Use in Patients of Advanced Age. JAMA Intern Med. 2019 Aug 1;179(8):1025-1033. doi: 10.1001/jamainternmed.2019.0631. PMID 31180477
- [Background] Zann V, McDermott J, Jacobs JW, Davidson JP, Lin F, Korner P, Blanks RC, Rosenbaum DP. Palatability and physical properties of potassium-binding resin RDX7675: comparison with sodium polystyrene sulfonate. Drug Des Devel Ther. 2017 Sep 6;11:2663-2673. doi: 10.2147/DDDT.S143461. eCollection 2017. PMID 28919716
- [Derived] Sondergaard H. Patient Involvement in the Design of an Innovative Clinical Study to Compare the Palatability of Anti-Hyperkalemia Medications. Patient Prefer Adherence. 2024 May 31;18:1059-1064. doi: 10.2147/PPA.S445399. eCollection 2024. PMID 38835400
- [Derived] Wheeler DC, Sondergaard H, Gwynn C, Hedman K, Hedberg J, Allum A, Chung HL, Nagard M, Stjernlof G, Wittbrodt E, Kim J, Morris J. Randomised, blinded, cross-over evaluation of the palatability of and preference for different potassium binders in participants with chronic hyperkalaemia in the USA, Canada and Europe: the APPETIZE study. BMJ Open. 2024 Feb 21;14(2):e074954. doi: 10.1136/bmjopen-2023-074954. PMID 38387989
- See also: AdSAM Emotional Response Modelling website. AdSAM Measure. — http://www.adsam.com/
- See also: Ingelfinger JR. A new era for the treatment of hyperkalemia? N Engl J Med [Internet]. 2015 Jan 15;372(3):275-7. — http://www.nejm.org/doi/10.1056/NEJMe1414112
- See also: Packham DK, Rasmussen HS, Lavin PT, El-Shahawy MA, Roger SD, Block G, et al. Sodium Zirconium Cyclosilicate in Hyperkalemia. N Engl J Med [Internet]. 2015;372(3):222-31. — http://www.nejm.org/doi/10.1056/NEJMoa1411487
- See also: Stokes JR, Boehm MW, Baier SK. Oral processing, texture and mouthfeel: From rheology to tribology and beyond. Curr Opin Colloid Interface Sci [Internet]. 2013;18(4):349-59. — http://dx.doi.org/10.1016/j.cocis.2013.04.010
- See also: Guinard JX, Mazzucchelli R. The sensory perception of texture and mouthfeel. Trends Food Sci Technol. 1996;7(7):213-9 — https://doi.org/10.1016/0924-2244(96)10025-X
- See also: CSR synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00016&attachmentIdentifier=2db63faf-57bf-4c0c-993c-e7cc29ef3ed7&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=